CLINICAL TRIAL: NCT01260688
Title: A Phase 2 Randomized Study of Cediranib (AZD2171) Alone Compared With the Combination of Cediranib (AZD2171) Plus BMS-354825 (Dasatinib, Sprycel) in Docetaxel Resistant, Castration Resistant Prostate Cancer
Brief Title: Cediranib Maleate With or Without Dasatinib in Patients With HRPC-Resistant to Treatment With Docetaxel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02544; PMH-PJC-002 (Other: University Health Network); PJC-002 (Other: Local protocol number); 8476 (Other: NIH protocol number); U01CA070095 (NIH); U01CA132123 (NIH); N01CM00071 (NIH)
Record Dates: First submitted 2010-12-14; First posted 2010-12-15 (Estimated); Results first posted 2013-12-05 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Hormone Refractory Prostate Cancer; Recurrent Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cediranib; Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Patients receive oral cediranib maleate once daily and oral dasatinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cediranib maleate; Drug: dasatinib
- Arm II (Experimental): Patients receive cediranib maleate as in arm I. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cediranib maleate

INTERVENTIONS:
Drug: cediranib maleate — Given orally
  Other Names: Recentin
Drug: dasatinib — Given orally
  Other Names: BMS-354825
  Arms: Arm I

SUMMARY:
This randomized phase II trial is studying the side effects and how well giving cediranib maleate together with or without dasatinib works in treating patients with hormone-resistant prostate cancer resistant to treatment with docetaxel. Cediranib maleate and dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth or by blocking blood flow to the tumor. It is not yet known whether giving cediranib maleate together with dasatinib or alone is an effective treatment for prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the progression-free survival of patients with docetaxel-resistant and castration-resistant prostate cancer treated with cediranib maleate with versus without dasatinib.

SECONDARY OBJECTIVES:

I. To confirm the safety and tolerability of cediranib maleate with versus without dasatinib in these patients.

II. To calculate objective response rates of cediranib maleate with versus without dasatinib, according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria, in patients with measurable disease at baseline.

III. To perform symptom assessment using the FACT-P questionnaire and the Present Pain Intensity (PPI) scale from the McGill-Melzack questionnaire.

IV. To explore bone resorption markers (e.g., c-telopeptide and bone alkaline phosphatase), and to correlate these biomarkers with clinical outcome.

OUTLINE: This is a multicenter study. Patients are stratified according to the presence of soft tissue (visceral or nodal) vs bone-only disease. Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive oral cediranib maleate once daily and oral dasatinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive cediranib maleate as in arm I. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed prostate cancer
* Measurable/non-measurable disease
* Prior hormonal therapy with medical LHRH agonist or orchiectomy castration (Castrate level of testosterone (< 50 ng/dL) required)
* Clinical/radiographic evidence of progression on or after docetaxel therapy
* No active pleural/pericardial effusion of any grade
* No meningeal metastases/untreated known brain metastases

  * Patients with treated brain metastasis with radiologic, clinical evidence of stability, with no evidence of cavitation/hemorrhage in the brain lesions allowed if asymptomatic and not requiring corticosteroids
* Life expectancy >3 months
* ECOG PS 0-2 (Karnofsky PS 60-100%)
* ANC >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 9 g/dL
* INR=< 1.3
* Total bilirubin =< 1.25 times ULN
* AST and ALT=< 2.0 times ULN (5 x ULN if clearly attributable to liver metastasis)
* Creatinine normal OR creatinine clearance >= 60 mL/min
* LVEF> institutional normal range by ECHO/MUGA
* Urine dipstick for protein < 1+ OR < 1 g on 24-hour urine collection

Exclusion Criteria:

* >5 years since any malignancy except in situ cancer, non-metastatic basal/squamous cell skin cancer, or other cancer for which the patient has been curatively treated
* Fertile patients must use effective contraception
* No condition that impairs ability to swallow/absorb
* No history of allergic reactions attributed to compounds of similar chemical/biologic composition to cediranib/dasatinib
* No systolic BP>150 mmHg and/or diastolic BP>100 mmHg
* QTc prolongation (>=480 msec by Fridericia correction) or other significant ECG abnormalities are ineligible
* No active/uncontrolled infections, serious illness, or medical conditions that would not permit patient to be managed according to protocol
* No known immunodeficiency syndrome
* No clinical/radiological evidence of severe/uncontrolled interstitial lung disease
* No history/concurrent idiopathic pulmonary fibrosis
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No unresolved toxicity>=CTCAE grade 2 (except alopecia) from prior anticancer therapy
* 4 weeks since prior anti-androgens
* 4 weeks since prior chemotherapy following docetaxel for metastatic disease (Any number of regimens allowed)
* 4 weeks since prior hormonal therapy or abiraterone
* 3 weeks since prior radioisotopes or radiotherapy and recovered
* No prior therapy with angiogenesis or Src or FAK inhibitors
* 3 weeks since prior major surgery and recovered
* 1 week since prior corticosteroids
* Concurrent zoledronic acid allowed provided patient has been receiving it prior to start of study treatment
* Concurrent medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of cediranib and dasatinib will be determined following review of their case by the principal investigator or co-investigator
* 14 days before and after study and no concurrent CYP3A4-active agents or substances (including strong inhibitors or inducers)
* Concurrent prophylactic low-dose warfarin (INR must be close monitored) or low-molecular weight heparin allowed
* No other concurrent investigational agents

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-10; Primary Completion 2013-01 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Hotte, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (8):
- United States (5):
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc - State Boulevard, Fort Wayne, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
- Canada (3):
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Spreafico A, Chi KN, Sridhar SS, Smith DC, Carducci MA, Kavsak P, Wong TS, Wang L, Ivy SP, Mukherjee SD, Kollmannsberger CK, Sukhai MA, Takebe N, Kamel-Reid S, Siu LL, Hotte SJ. A randomized phase II study of cediranib alone versus cediranib in combination with dasatinib in docetaxel resistant, castration resistant prostate cancer patients. Invest New Drugs. 2014 Oct;32(5):1005-16. doi: 10.1007/s10637-014-0106-5. Epub 2014 May 3. PMID 24788563

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was open to recruitment on October 25, 2010 and closed to accrual on July 31, 2012. Study participants were identified in clinic. The target enrolment was 50 study participants; however only 22 participants enrolled as the study was terminated due to discontinuation of cediranib drug supply due to clinical development discontinuation.
Groups:
- Arm I - Cediranib Plus Dasatinib: Patients receive oral cediranib maleate once daily and oral dasatinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Arm II - Cediranib Alone: Patients receive cediranib maleate as in arm I. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm I - Cediranib Plus Dasatinib | Arm II - Cediranib Alone
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I - Cediranib Plus Dasatinib | Arm II - Cediranib Alone | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 9 | 10 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (7.1) | 72.7 (6.5) | 69 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 11 | 11 | 22
Region of Enrollment [Number; unit: participants]
  Canada | 9 | 8 | 17
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: 12-week Progression-free Survival as Per the Prostate Cancer Clinical Trials Working Group (PCWG2)
Description: Progression is defined using the Prostate Cancer Clinical Trials Working Group (PCWG2) criteria, which includes a compilation of prostate-specific antigen (PSA), bone scan, and CT-scan assessments (Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 3 months
Population: All patients were included in the analysis for 12-week PFS.
Measure: Number; unit: participants
Groups:
- Arm II - Cediranib Alone: Patients receive oral cediranib maleate once daily for 28 days. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm I - Cediranib Plus Dasatinib | Arm II - Cediranib Alone
Number analyzed (Participants) | 11 | 11
participants | 2 | 8

2. Secondary Outcome: Number of Participants With Toxicities
Description: Incidence of toxicities graded according to the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) v4.0
Time Frame: Up to 30 days after last dose of study drugs
Measure: Number; unit: participants
Groups:
- Arm I - Cediranib Plus Dasatinib: Patients receive oral cediranib maleate (20mg) once daily and oral dasatinib (100mg) once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity
- Arm II - Cediranib Alone: Patients receive oral cediranib maleate (20mg) once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity
Arm/Group | Arm I - Cediranib Plus Dasatinib | Arm II - Cediranib Alone
Number analyzed (Participants) | 11 | 11
participants | 11 | 11

3. Secondary Outcome: Qualtiy of Life Assessment Number of Participants With a Score ≥2 on the Present Pain Intensity (PPI) Scale
Description: Present Pain Intensity (PPI) scale. Scale is measured 0-5, where 0=no pain, 1=mild pain, 2=discomforting pain, 3=distressing pain, 4=horrible pain and 5=excruciating pain Participants who were up to completing the assessment (did not decline) and who reported a score >=2 at the end of any cycle are reported.
Time Frame: After every cycle (median duration on study = 4 cycles)
Population: Analysis was performed patients receiving single agent cediranib or combination of cediranib plus dasatinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I - Cediranib Plus Dasatinib | Arm II - Cediranib Alone
Number analyzed (Participants) | 11 | 11
Participants | 4 | 8

4. Secondary Outcome: Number Who Experienced Study Medication Dose Intensity
Description: Number of patients who experienced study medication dose of over 80% during Cycle 1 was assessed.
Time Frame: Cycle 1 (an average of 28 days)
Measure: Number; unit: participant
Arm/Group | Arm I - Cediranib Plus Dasatinib | Arm II - Cediranib Alone
Number analyzed (Participants) | 11 | 11
participant | 6 | 9

5. Secondary Outcome: Treatment Discontinuation
Description: Discontinuation of treatment in cycle 1 (average of 28 days)
Time Frame: Cycle 1 (average of 28 days)
Population: Analysis was performed on study participants enrolled on the trial assessing number of patients who discontinued treatment in cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I - Cediranib Plus Dasatinib | Arm II - Cediranib Alone
Number analyzed (Participants) | 11 | 11
Participants | 7 | 6

6. Secondary Outcome: Treatment Discontinuation Due to Adverse Events (AEs)
Description: Treatment discontinuation due to Adverse Events
Time Frame: Through study completion (median duration on study = 4 cycles)
Measure: Number; unit: participants
Arm/Group | Arm I - Cediranib Plus Dasatinib | Arm II - Cediranib Alone
Number analyzed (Participants) | 11 | 11
participants | 2 | 1

7. Secondary Outcome: Non-AE Related Treatment Discontinuation
Description: Non-Adverse Event related Treatment Discontinuation
Time Frame: Through study completion (median duration on study = 4 cycles)
Measure: Number; unit: participants
Arm/Group | Arm I - Cediranib Plus Dasatinib | Arm II - Cediranib Alone
Number analyzed (Participants) | 11 | 11
participants
  Progressive Disease | 4 | 4
  Death | 0 | 2
  Other | 5 | 4

8. Secondary Outcome: Overall Response Rate
Description: Best overall response rate of each evaluable patient
Time Frame: Duration of Study (median duration on study = 4 cycles)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I - Cediranib Plus Dasatinib | Arm II - Cediranib Alone
Number analyzed (Participants) | 11 | 11
months | 2.6 [1.4 to NA] — confidence interval not reached. | 6.4 [1.9 to NA] — confidence interval not reached.

9. Secondary Outcome: Treatment Related Deaths
Description: Number of treatment related deaths
Time Frame: Through study completion (median duration on study = 4 cycles)
Population: In Arm II (Cediranib alone), 1 patient presented retroperitoneal hemorrhage (Grade 5).
Measure: Number; unit: participants
Arm/Group | Arm I - Cediranib Plus Dasatinib | Arm II - Cediranib Alone
Number analyzed (Participants) | 11 | 11
participants | 0 | 1

10. Secondary Outcome: Participants for Which Bone Biomarkers for Beta-C Telopeptide Was Reduced
Description: Participants for which beta-C telopeptide was reduced
Time Frame: Through study completion (median duration on study = 4 cycles)
Population: Analysis was done on study participatns for which beta-C telopeptide was reduced.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I - Cediranib Plus Dasatinib | Arm II - Cediranib Alone
Number analyzed (Participants) | 11 | 9
Participants | 7 | 6

11. Secondary Outcome: Number of Participants With Increased Alkaline Phosphatase BAP
Description: Number of participants with increased alkaline phosphatase BAP
Time Frame: Through study completion (median duration on study = 4 cycles)
Measure: Number; unit: participants
Arm/Group | Arm I - Cediranib Plus Dasatinib | Arm II - Cediranib Alone
Number analyzed (Participants) | 9 | 11
participants | 5 | 10

12. Secondary Outcome: Dose Interruption Due to AEs
Description: The number of participants with dose-interruptions in each arm due to adverse events
Time Frame: Through study completion (median duration on study = 4 cycles)
Population: Analysis was performed on study participants assessing the number of participants with dose-interruptions due to adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I - Cediranib Plus Dasatinib | Arm II - Cediranib Alone
Number analyzed (Participants) | 11 | 11
Participants | 8 | 6

13. Secondary Outcome: Dose Reductions
Description: The number of participants with dose reductions in each arm
Time Frame: Duration of Study (median duration on study = 4 cycles)
Population: Analysis conducted on the number of participants with dose reductions in each arm of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I - Cediranib Plus Dasatinib | Arm II - Cediranib Alone
Number analyzed (Participants) | 11 | 11
Participants | 5 | 4

14. Secondary Outcome: Overall Response Rate
Description: Response Rate of Stable Disease and Progressive Disease
Time Frame: Duration of Study (median duration on study = 4 cycles)
Population: Analysis of number of participants who experienced response rates of SD and PD.
Measure: Number; unit: percentage of participants
Arm/Group | Arm I - Cediranib Plus Dasatinib | Arm II - Cediranib Alone
Number analyzed (Participants) | 11 | 11
percentage of participants
  Stable Disease | 22 | 77
  Progressive Disease | 45 | 18

15. Secondary Outcome: Quality of Life Assessment Using Functional Assessment of Cancer Therapy - Prostate (FACT-P) Questionnaire
Description: Scale is measured on a range from 0 (worst quality of life) to 156 (best quality of life).
Time Frame: Up to 16 weeks
Population: Some participants (overall and post-baseline) did not complete the questionnaire or failed to answer more than 7 questions and could not be included in the analysis (a summary score could not be calculated).
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Arm I - Cediranib Plus Dasatinib | Arm II - Cediranib Alone
Number analyzed (Participants) | 10 | 10
units on a scale
  Baseline | 117.5 [78.3 to 129.5] | 108.5 [83 to 124]
  Cycle 2 (8 weeks): number analyzed (Participants) | 8 | 8
  Cycle 2 (8 weeks) | 120.6 [74 to 131.5] | 107 [67 to 131]
  Cycle 3 (12 weeks): number analyzed (Participants) | 8 | 5
  Cycle 3 (12 weeks) | 109.1 [70.2 to 132] | 105.8 [91 to 119]
  Cycle 4 (16 weeks): number analyzed (Participants) | 5 | 2
  Cycle 4 (16 weeks) | 114.5 [67.5 to 119] | 93.8 [93.7 to 94]

ADVERSE EVENTS:
Arm/Group | Arm I - Cediranib Plus Dasatinib | Arm II - Cediranib Alone
Serious Adverse Events (participants affected / at risk) | 5/11 | 7/11
Other Adverse Events (participants affected / at risk) | 11/11 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Cediranib Plus Dasatinib (N=11) | Arm II - Cediranib Alone (N=11)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bile obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2)
Pending Spinal Cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) — In Arm II (Cediranib alone), 1 patient presented retroperitoneal hemorrhage (Grade 5)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I - Cediranib Plus Dasatinib (N=11) | Arm II - Cediranib Alone (N=11)
Hypertension (Vascular disorders) | 9 | 11
Anemia (Blood and lymphatic system disorders) | 11 | 11
Diarrhea (Gastrointestinal disorders) | 8 | 7
Fatigue (General disorders) | 11 | 9
Alkaline Phosphatase Increased (Investigations) | 8 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Lymphocyte Count decreased (Investigations) | 8 | 9
Nausea (Gastrointestinal disorders) | 6 | 4
Peripheral Sensory Neuropathy (Nervous system disorders) | 6 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 3
Hematuria (Renal and urinary disorders) | 2 | 5
Obesity (Metabolism and nutrition disorders) | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 5 | 6
Anxiety (Psychiatric disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 5 | 7
Weight loss (Investigations) | 9 | 4
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 3
Platelet Count Decreased (Investigations) | 5 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Electrocardiogram QT Corrected Interval Prolonged (Investigations) | 2 | 4
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hot Flashes (Vascular disorders) | 4 | 2
Depression (Psychiatric disorders) | 3 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 8
Sinus tachycardia (Cardiac disorders) | 1 | 3
Urinary incontinence (Renal and urinary disorders) | 1 | 4
Hyponatremia (Metabolism and nutrition disorders) | 5 | 6
Edema limbs (General disorders) | 2 | 5
Stomach pain (Gastrointestinal disorders) | 1 | 1
Aspartate aminotransferase Increase (Investigations) | 8 | 4
Insomnia (Psychiatric disorders) | 1 | 4
Proteinuria (Renal and urinary disorders) | 4 | 6
Dysgeusia (Nervous system disorders) | 2 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 7
Creatinine increased (Investigations) | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 3
Alanine Aminotransferase Increased (Investigations) | 2 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Sinus bradycardia (Cardiac disorders) | 0 | 2
Urinary frequency (Renal and urinary disorders) | 4 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 5 | 3
Oral dysesthesia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Erythrocytes decreased (Investigations) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 2
Scalp dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 2
Flatulence (Gastrointestinal disorders) | 1 | 1
Hypothyroidism (Endocrine disorders) | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Seizure (Nervous system disorders) | 0 | 1
Bloating (Gastrointestinal disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 4 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
White blood cell decreased (Investigations) | 1 | 2
Cholesterol high (Investigations) | 0 | 1
Diminished breath sounds (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Fecal incontinence (Gastrointestinal disorders) | 0 | 1
Genital edema (Reproductive system and breast disorders) | 0 | 1
Headache (Nervous system disorders) | 4 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 2
Restless legs (Musculoskeletal and connective tissue disorders) | 0 | 1
Bilateral rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chills (General disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Dizziness (Nervous system disorders) | 3 | 2
Fever (General disorders) | 2 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Irregular heart rate and rhythm (Cardiac disorders) | 0 | 1
Lymphocyte count increased (Investigations) | 0 | 1
Nocturia (Renal and urinary disorders) | 1 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 2
rectal hemorrhage (Gastrointestinal disorders) | 1 | 1
Spasticity (Nervous system disorders) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Blood bilirubin increased (Musculoskeletal and connective tissue disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1
Disease Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Glucose Intolerance (Metabolism and nutrition disorders) | 2 | 1
hemorrhoidal hemorhage (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Lung infection (Infections and infestations) | 1 | 1
Mucositis oral (Gastrointestinal disorders) | 4 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Neutrophil Count decreased (Investigations) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Retroperitoneal hemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1
Serum amylase increased (Investigations) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 6 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0
Hearing impaired (Ear and labyrinth disorders) | 2 | 0
Ventricular Diastolic disorder (Cardiac disorders) | 1 | 0
Dry throat (Gastrointestinal disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Osteonecrosis of Jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Blood in stool (Gastrointestinal disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Lip sore (Gastrointestinal disorders) | 1 | 0
Low T3 (Investigations) | 1 | 0
Movements involuntary (Musculoskeletal and connective tissue disorders) | 1 | 0
Rib pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Sore throat (Gastrointestinal disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Gastroparesis (Gastrointestinal disorders) | 1 | 0
Low T4 (Investigations) | 1 | 0
Lower Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Mucosal infection (Infections and infestations) | 1 | 0
Palmar-Plantar Erythrodysesthesia (Skin and subcutaneous tissue disorders) | 1 | 0
Runny nose (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Clinical development discontinuation of Cediranib leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less